CLINICAL TRIAL: NCT06008847
Title: Capsule Endoscopy Delivery at sCale Through Enhanced AI anaLysis Study
Acronym: CESCAIL
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: RA545021
Record Dates: First submitted 2022-04-07; First posted 2023-08-24 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Bowel Cancer
Keywords: bowel; cancer; AI
MeSH Terms: conditions — Intestinal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Gastrointestinal Symptoms: Participant aged over 18 with referred lower gastrointestinal symptoms

SUMMARY:
The CESCAIL study tests the use of Artificial Intelligence (AI) on a video taken from a minimally-invasive imaging device, to improve efficiency and accuracy of the detection of polyps, which are little outgrowths within the lining of the bowel.

DETAILED DESCRIPTION:
Participants will be continuing to follow their standard care pathway, and there are no additional requirements of the participants other than providing consent for their pseudonymised capsule video and data to be used to test the AI system.

The participant's final diagnosis will only be determined by the clinician's standard analysis pathway and not influenced by the AI enabled analysis pathway. All data is de-identified before a video is created and re-identified only once the standard final report is signed-off by the referring clinician. Therefore, the risk of patient harm due to exposed data is minimised.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Patients who have been selected by overseeing clinician meeting NHS England criteria to undergo colon capsule endoscopy as part of their standard of care

Exclusion Criteria:

* Patients unable to provide consent to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, aged 18 and over
Sampling Method: Non-Probability Sample
Enrollment: 674 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of polyp detection in AI enabled CCE reporting | 11 months
  Sensitivity and specificity of polyp detection in AI enabled CCE reporting
Time taken to read video by clinicians and AI tool | 11 months
  Time taken to read video by clinicians and AI tool

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry and Warwickshire, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No